CLINICAL TRIAL: NCT00000260
Title: Effects of Behavioral Contingencies on Effects of Nitrous Oxide
Brief Title: Effects of Behavioral Contingencies on Effects of Nitrous Oxide - 12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: NIDA-08391-12; R01DA008391 (NIH); R01-08391-12
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Opioid-Related Disorders; Substance-Related Disorders
Keywords: nitrous oxide; subjective effects; reinforcer; inhalant; healthy volunteer
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders | interventions — Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous oxide

SUMMARY:
The purpose of this study is to conduct experiments to examine subjective and reinforcing effects of nitrous oxide. Mood altering and psychomotor effects will be tested on non-drug abusers and preference procedures will be used to assess reinforcing effects. Comparisons between nitrous oxide, opiates, and benzodiazepine antagonists will be made. To examine the effects of different behavioral contingencies in modulating the reinforcing effects of nitrous oxide in healthy volunteers.

ELIGIBILITY:
Please contact site for information.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1997-06; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Mood
Choice of nitrous oxide vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: James Zacny, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Anesthesia & Critical Care, Chicago, Illinois, United States